CLINICAL TRIAL: NCT02509832
Title: COOL-AMI EU PILOT TRIAL: A Multicenter, Prospective, Randomized Controlled Trial To Assess Cooling as an Adjunctive Therapy to Percutaneous Intervention in Patients With ACUTE MYOCARDIAL INFARCTION
Brief Title: COOL AMI EU Pilot Trial to Assess Cooling as an Adjunctive Therapy to Percutaneous Intervention in Patients With Acute Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZOLL Circulation, Inc., USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EDC-2420
Record Dates: First submitted 2015-07-24; First posted 2015-07-28 (Estimated); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Acute Myocardial Infarction
Keywords: Therapeutic Hypothermia (TH); Acute Myocardial Infarction (AMI); Percutaneous Coronary Intervention (PCI)
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cooling + PCI (Other): The subjects will be considered to be enrolled in the Test Arm of the trial when all inclusion and exclusion criteria have been met, the informed consent form has been signed, and randomization to the Test Arm of the trial to allow cooling with the Proteus IVTM System before and after PCI.
  Interventions: Device: Cooling + PCI
- PCI only (Other): The subjects will be considered to be enrolled in the Control Arm of the trial when all inclusion and exclusion criteria have been met, the informed consent form has been signed, and randomization to the Control Arm of the trial to allow PCI only.
  Interventions: Device: PCI only

INTERVENTIONS:
Device: Cooling + PCI — Cooling with ZOLL Proteus IVTM System before and after Percutaneous Coronary Intervention (PCI)
  Arms: Cooling + PCI
Device: PCI only — Standard of Care for PCI
  Arms: PCI only

SUMMARY:
COOL AMI EU Pilot Trial: A Multicenter, Prospective, Randomized Controlled Trial to Assess Cooling as an adjunctive Therapy to Percutaneous Intervention in Patients with Acute Myocardial Infarction.

Evaluate the retention of subjects after integrating therapeutic hypothermia using the ZOLL Proteus IVTM System into existing STEMI treatment protocols for subjects who present with acute anterior myocardial infarction.

DETAILED DESCRIPTION:
Evaluate the retention of subjects after integrating therapeutic hypothermia using the ZOLL Proteus IVTM System into existing STEMI treatment protocols for subjects who present with acute anterior myocardial infarction.

ELIGIBILITY:
All Inclusion Criteria must be answered YES for subject to be eligible for trial Inclusion Criteria:

1. ≥ 18 years of age.
2. symptoms consistent with AMI (chest pain, unresponsive to nitroglycerin, ≥ 30 minutes and < 6 hours.
3. Anterior MI with ST-segment elevation of 0.2 mV in two or more anterior contiguous precordial leads.
4. Eligible for PCI.
5. Opportunity for at least 10 minutes of cooling with the Proteus IVTM System prior to PCI.
6. Written, informed consent to participate in this clinical trial.

Exclusion Criteria:

All Exclusion Criteria must be answered NO for subject to be eligible for trial inclusion.

1. Previous myocardial infarction.
2. Cardiogenic shock (systolic blood pressure [SBP] <80 mmHg and non-responsive to fluids, or SBP <100 mmHg with vasopressors, or requirement for an intra-aortic balloon pump [IABP]).
3. Resuscitated cardiac arrest, atrial fibrillation, or Killip risk stratification class II through IV
4. Aortic dissection or requires an immediate surgical or procedural intervention other than PCI
5. Congestive Heart Failure (CHF), hepatic failure, end- stage kidney disease or severe renal failure (clearance < 30ml/min/1.73m2).
6. Fever (temperature > 37.5 °C) or infection with fever in the last 5 days.
7. Previous CABG.
8. Stroke within 90 days of admission.
9. Cardio-pulmonary decompensation present or imminent
10. Contraindications to hypothermia, such as patients with known hematologic dyscrasias which affect thrombosis (e.g., cryoglobulinemia, sickle cell disease, serum cold agglutinins) or vasospastic disorders (such as Raynaud's or thromboangitis obliterans)
11. Hypersensitivity or contraindication to aspirin, heparin, or sensitivity to contrast media, which cannot be adequately pre-medicated.
12. History of bleeding diathesis, coagulopathy, cryoglobulinemia, sickle cell anemia, or will refuse blood transfusions.
13. Height of <1.5 meters (4 feet 11 inches).
14. Hypersensitivity to buspirone hydrochloride or Pethidine (Meperidine) and/or treatment with a monoamine oxidase inhibitor in the past 14 days.
15. History of severe hepatic or renal impairment, untreated hypothyroidism, Addison's disease, benign prostatic hypertrophy, or urethral stricture that in the opinion of the physician would be incompatible with Pethidine administration.
16. Inferior Vena Cava filter in place (IVC).
17. The patient has a pre-MI life expectancy of <1 year due to underlying medical conditions or pre-existing co-morbidities.
18. Known, unresolved history of drug use or alcohol dependency, or lacks the ability to comprehend or follow instructions.
19. Currently enrolled in another investigational drug or device trial that has not completed the primary endpoint.
20. Apprehension or unwilling to undergo the required MRI imaging at follow-up, has a documented or suspected diagnosis of claustrophobia, or has Gadolinium allergy
21. Received thrombolytic therapy en route to the hospital
22. Clinical evidence of spontaneous reperfusion as observed symptomatically and/ or from ECG findings (partial or complete ST resolution in ECG before randomization) upon admission
23. Vulnerable subject, for instance, a person in detention (i.e., prisoner or ward of the state)
24. Female who is known to be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-07; Primary Completion 2018-03 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Proportion of all subjects who complete the follow-up and cMR imaging requirements at 30-day follow up period | 30 day

SECONDARY OUTCOMES:
1. Anterior Infarct Size (IS) as assessed by Cardiac Magnetic Resonance (cMR) at 4 - 6 days following the index procedure for subjects in Test and Control Arms | 4 - 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Holzer, Principal Investigator — Universitätsklinik für Notfallmedizin Allgemeines Krankenhaus der Stadt Wien; Marko Noc, Principal Investigator — University Medical Center Ljubljana Slovenia
Locations (13):
- Universitätsklinik für Notfallmedizin Allgemeines Krankenhaus der Stadt Wien, Vienna, Austria
- North Estonia Medical Center, Tallinn, Estonia
- Hungary (3):
  - Heart Center Balatonfüred, Balatonfüred
  - Medical and Health Science Center University of Debrecen, Debrecen
  - Heart Institute University of Pecs, Pécs
- Poland (3):
  - Medical University in Łódź, Bieganski Hospital, Lodz
  - National Institute of Cardiology, Department of Interventional Cardiology & Angiology, Warsaw
  - Silesian Center for Heart Diseases, Zabrze
- Serbia (2):
  - Clinical Center of Serbia Head of Department for invasive diagnostics (Division of Cardiology), Belgrade
  - University Clinical Hospital Center Zemun, Zemun
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- Skane University Hospital Lund University, Lund, Sweden
- Essex Cardiothoracic Centre, Anglia Ruskin University, Basildon, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided